CLINICAL TRIAL: NCT07395414
Title: Randomized Cross-over Study
Brief Title: Effect of Different Work-to-rest Ratios During Simulated Taekwondo Combat on Blood Lactate, Heart Rate and Perceptual Responses in Elite Taekwondo Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, Bayram Ceylan, Assoc. Prof., Kastamonu University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2022-KAEK-12
Record Dates: First submitted 2026-01-24; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: HIIT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Visit 1 (Experimental)
  Interventions: Other: Free combat
- Visit 2 (Experimental)
  Interventions: Other: 1:2 work to rest ratio
- Visit 3 (Experimental)
  Interventions: Other: 2:1 work to rest ratio

INTERVENTIONS:
Other: Free combat — Athletes completed a taekwondo combat for 3 sets of 2 minutes
  Arms: Visit 1
Other: 1:2 work to rest ratio — Athletes completed a taekwondo combat for 3 sets of 2 mins with 1:2 work to rest ratio (10 sec work and 20 sec rest)
  Arms: Visit 2
Other: 2:1 work to rest ratio — Athletes completed a taekwondo combat for 3 sets of 2 minutes with 2:1 work to rest ratio (20 second work and 10 second rest)
  Arms: Visit 3

SUMMARY:
This randomized cross-over study measured physiological and perceptual responses of taekwondo athletes following a free combat and combats with different W:R ratios. This study was carried out with 4 visits. The first one included body composition measurements and familiarization to the sessions and measurements. During the rest 3 visit, athletes performed simulated combats free and with 1:2 (10 sec work and 20 sec rest), and 2:1 (20 sec work and 10 sec rest) W:R ratios. During all combat sessions, athletes heart rate (HR), blood lactate (bLA), and counter-movement jump performance (CMJ) were measured at rest and at the end of each combat. HR was also measured following each set. Athletes' rating of perceived exertion (RPE) and perceived muscle soreness (PMS) were measured immediately after each combat.

ELIGIBILITY:
Inclusion Criteria:

* having at least brown belt,
* having at least 5 years of taekwondo experience,
* having no injuries for the last 6 months that prevent participating to trainings,
* competing at national championship and international tournaments during the last year

Exclusion Criteria:

* not having a brown belt,
* having less than 5 years of taekwondo experience,
* having injuries for the last 6 months that prevent participating to trainings,
* Not competing at national championship and international tournaments during the last year

Ages: 18 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-05 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
Lactate | Immediately after each intervention
  Athletes' lactate levels immediately after the exercise
Heart rate | Before and immediately after each intervention
  Athletes' heart rate responses
CMJ | Before and immediately after each intervention
  Athletes' CMJ was measured before and after each exercise session.

SECONDARY OUTCOMES:
RPE | Immediately after each intervention
  Athletes' RPE was measured immediately after each exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Bayram Ceylan, PhD, Principal Investigator — Kastamonu University
Locations (1):
- Kastamonu University Faculty of Sport Sciences Physiology Lab, Kastamonu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bridge CA, Jones MA, and Drust B. Physiological responses and perceived exertion during international Taekwondo competition. International Journal of Sports Physiology And Performance 4: 485-493, 2009.
- [Background] Bouhlel E, Jouini A, Gmada N, Nefzi A, Ben Abdallah K, and Tabka Z. Heart rate and blood lactate responses during Taekwondo training and competition. Science & Sports 21: 285-290, 2006.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/14/NCT07395414/Prot_SAP_000.pdf